CLINICAL TRIAL: NCT06738108
Title: Safety and Effectiveness of EKOS in PE Patients
Brief Title: EKOS in Patients With Pulmonary Embolism (PE)
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, Lecturer of clinical pharmacy, Beni-Suef University
Other Study IDs: ECOSII
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Embolism
Keywords: ECOS
MeSH Terms: conditions — Pulmonary Embolism | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECOS group: ECOS
  Interventions: Drug: ECOS
- Control group: IV infusion tpa
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: ECOS — The EkoSonic Endovascular System, developed by EKOS Corporation, is a specialized CDT system that combines ultrasound technology with thrombolytic infusion to treat PE
  Groups: ECOS group
Drug: Control group — Alteplase IV infusion
  Other Names: IV alteplase infusion
  Groups: Control group

SUMMARY:
A retrospective cohort study assessed patients who underwent EKOS intervention following the failure of initial therapeutic anticoagulation for managing acute pulmonary embolism at a tertiary hospital.

DETAILED DESCRIPTION:
A retrospective cohort study assessed patients who underwent EKOS intervention following the failure of initial therapeutic anticoagulation for managing acute pulmonary embolism at a tertiary hospital. Patients aged at least 18 years with a diagnosis of submassive or massive acute PE were included. Patients were excluded if they either did not receive EKOS intervention or were presented with stable PE. The primary outcome was the change in RV/LV diameter ratio from baseline to first outpatient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years diagnosed with massive or submassive acute PE.

Exclusion Criteria:

1. Patients presented with stable PE
2. Patients did not receive EKOS intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Submassive PE was defined as having right ventricular (RV) dysfunction: detected via CT scan or echocardiography, with signs such as RV enlargement, RV hypokinesis, or RV/LV ratio >0.9 to 1.0), elevated cardiac biomarkers like troponin or BNP, which indicate strain or injury to the heart muscle with a maintained blood pressure (SBP equal to or > 90 mm Hg with no signs of shock.
  Massive PE was defined as SBP <90 mm Hg for at least 15 minutes or require vasopressors to maintain adequate blood pressure with clinical signs of poor perfusion, including altered mental status, cool extremities, low urine output, or sudden loss of heart function due to obstructed blood flow from the pulmonary artery.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
The change in RV/LV diameter ratio | one month
  The change in RV/LV diameter ratio from baseline to first outpatient follow-up as documented on an echocardiogram.

SECONDARY OUTCOMES:
All-cause 30-day readmission | one month
  All-cause 30-day readmission

CONTACTS AND LOCATIONS:
Locations (1):
- Saudi German Hospital, Cairo, Egypt